CLINICAL TRIAL: NCT02454790
Title: Standard Follow-up Program (SFP) for Esophageal Cancer Patients Treated With Radiotherapy or Chemoradiation
Brief Title: Standard Follow-Up Program (SFP) for Patients With Esophageal Cancer
Acronym: SFP OES
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: SFP OES
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Esophageal Cancer
Keywords: Acute toxicity; Late toxicity; Prediction models
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy; Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Radiotherapy
  Other Names: Chemoradiation

SUMMARY:
Motive:

In order to improve the treatment technique, a comprehensive follow-up program is needed to obtain all relevant patient, treatment and toxicity data from esophageal cancer patients.

Goal:

To set-up and maintain a database containing treatment results in terms of tumor control, side effects, complications and patient-reported quality of life.

A standard database of patients receiving photon treatment will be created. These data are then linked to dose-volume data of radiotherapy, with the aim to build prediction models for both tumor control and toxicity after radio (chemo) therapy that can later be used for selecting patients for proton treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with esophageal cancer
* Patients receiving a radiotherapy dose > 40 Gy

Exclusion Criteria:

* Failure to comply with any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer receiving a radiotherapy dose > 40 Gy
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-09; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | Highest during and within 2 weeks after last day of radiation therapy
Late toxicity | Highest within one year after last day of radiation therapy

SECONDARY OUTCOMES:
Overall survival | At 1,2,3,4 and 5 years after first day of radiation therapy
Loco-regional tumor control | At 1,2,3,4 and 5 years after first day of radiation therapy

OTHER OUTCOMES:
Patient-rated symptoms and Quality-of-Life | Before first day of radiation therapy and at 3,6,12,24,36,48,60 months after first day of radiation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands